CLINICAL TRIAL: NCT06013280
Title: The Effect of Relaxation and Breathing Exercise on Post-Earthquake Stress Related Symptoms
Brief Title: The Effect of Relaxation Techniques on Earthquake Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, sabiha sancaktar, Research Assistant, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulMUH-FTR-SIS-01
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Earthquake; Mental Health Issue
Keywords: earthquake; physiotherapy; breathing exercise; relaxing exercise; stress; mental health
MeSH Terms: conditions — Psychological Well-Being | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Two groups with a control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxing Exercise Group (Experimental): Relaxing exercise group participants applied 40 minutes of progressive muscle relaxation and breathing exercises, 3 times a week for 4 weeks
  Interventions: Other: Progresive Muscle Relaxation and Breathing Exercise
- Control Group (No Intervention): This group received no intervention, continued their daily life as usual.

INTERVENTIONS:
Other: Progresive Muscle Relaxation and Breathing Exercise — Intervention protocol contains 40 minuntes sessions, which involved tensing and relaxing the body along with deep breathing.
  Protocol consisted with; Warm-up (5 minutes breathing exercise) Progressive Muscle Relaxation Exercises (The participants performed PMR for each body part in a particular order, beginning with the face muscles and head, followed by neck, shoulders, chest, abdomen, legs, and feet. This muscle tensing and relaxing procedures were performed in accompaniment with deep breathing.) Cool-down (5 minutes breathing exercise)
  Arms: Relaxing Exercise Group

SUMMARY:
The aim of this study is to investigate the effect of relaxation and breathing exercises on individuals experiencing post-earthquake stress-related symptoms.

DETAILED DESCRIPTION:
Earthquakes negatively affect survivors both physically and psychologically. Early psychological symptoms after disasters are considered normal responses to an abnormal event. Therefore, it is not unexpected to feel very intense negative emotions after such traumas. However, the chronicity of these negative emotions puts the lives of individuals at risk. Mental problems such as stress, depression, posttraumatic stress disorder and anxiety are seen at high levels among earthquake survivors. In this study, it was aimed to investigate the effect of relaxation and breathing exercises applied to earthquake survivors who experienced post-earthquake stress-related symptoms.

There are two gropus: relaxing exercise group and control group. Relaxing and breathing exercise protocol is only for relaxing exercise group. A protocol consisting of 40 minutes of progressive muscle relaxation exercise and breathing exercises, 3 times a week for 4 weeks, was planned. Control group participants were asked to continue their daily lives. Evaluations were made before and 4 weeks after the intervention and stress-related symptoms were measured.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a Beck anxiety inventory score greater than 8 and anxiety experience for more than 1 month
* Individuals who experienced the earthquake of February 6, 2023 Kahramanmaraş / Türkiye and agreed to participate in the study
* Individuals without cognitive impairment
* Individuals who can understand and apply verbal commands in Turkish

Exclusion Criteria:

* Any history of psychiatric medication support for the last 6 months
* Any history of psychological problems before the earthquake

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety (BAI) | four weeks
  Beck Anxiety Inventory is a brief measure of anxiety with a focus on somatic symptoms of anxiety that was developed as a measure adept at discriminating between anxiety and depression. It is a self-report scale consisting of 21 items. Respondents indicate how much they have been bothered by each symptom over the past week. Responses are rated on a 4-point Likert scale and range from 0 (not at all) to 3 (severely). The total score ranges from 0-63. The following guidelines are recommended for the interpretation of scores: 0-9, normal or no anxiety; 10-18, mild to moderate anxiety; 19-29, moderate to severe anxiety; and 30-63, severe anxiety.

SECONDARY OUTCOMES:
The Posttraumatic Stress Diagnostic Scale (PDS) | four weeks
  The Posttraumatic Stress Diagnostic Scale (PDS) is a 49-item self-report questionnaire designed to measure the severity of PTSD symptoms. A total score of 1-10 is considered as mild symptoms 11-20 moderate symptoms 21-35 as moderate to severe symptoms and 36 or over as is considered to reflect severe symptoms.
Beck Depression Inventory (BDI) | four weeks
  The Beck Depression Inventory Second is a 21-item self-report instrument measuring the existence and severity of symptoms of depression.
Perceived Stress Scale -10 | four weeks
  The Perceived Stress Scale (PSS-10) is a widely used and well validated 10 item self report questionnaire designed to measure to what degree the respondent appraises his life situation over the past month. A higher score is associated with greater vulnerability.
Pittsburgh Sleep Quality Index | four weeks
  This scale contains seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efciency, sleep disturbances, use of sleep medication, and daytime dysfunction. There are 19 questions in this questionnaire, with a total score ranging from 0-21. A higher score indicates worse sleep quality.
SF-12 | four weeks
  SF-12 evaluates health - related quality of life.It was developed to shorten the SF-36 using a regression method. As per the dimensionality of the SF-36, SF-12 encompasses 12 items that have to be scored in two 0-100 components: the physical component summary (PCS12) and the mental component summary (MCS12). SF-12 items are referred to as physical restrictions, physical functioning, bodily pain, general health compared with others, vitality, social functioning, role limitations due to emotional issues, and mental health (MH). Higher scores indicates higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Irem Sancaktar, M.Sc., Principal Investigator — Istanbul Medipol Hospital
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)